CLINICAL TRIAL: NCT06751160
Title: Comparative Effects of Dry Needling Versus Soft Tissue Mobilization on Hamstring Tightness in Chronic Low Back Pain
Brief Title: Comparative Effects of Dry Needling Versus Soft Tissue Mobilization on Hamstring Tightness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0106
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hamstring Tightness; Chronic Low-back Pain
Keywords: Chronic Low Back Pain; Disability; Dry Needling; Hamstring Tightness; Soft Tissue Mobilization
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): Dry Needling along with baseline treatment
  Interventions: Other: Dry Needling
- Soft Tissue Mobilization (Experimental): Soft Tissue Mobilization along with baseline treatment
  Interventions: Other: Soft Tissue Mobilization

INTERVENTIONS:
Other: Dry Needling — Baseline Treatment: Hot pack will be applied for 15 minutes on Hamstrings and lower back and transcutaneous electrical nerve stimulation (TENS) at lower back for warm up and pain relief to both groups. Then spinal mobilization (Poster lateral glide) of grade 1 and 2 (3 sets of 6 repetitions) i.e. within the spine resistance.
  Dry Needling will be given to group A along with baseline treatment through following protocol:
  Patient will be in prone lying. Sterilized disposable dry needles of 0.25*60mm will be used. Dry needling will be performed on three points on Hamstring muscle for one minute each. We considered a line between ischial tuberosity and head of fibula to target long head of bicep femoris (60% of line) and short head of bicep femoris (30% of line). Semitendinosus and Semi Membranosus were targeted at a point of 60% of line from ischial tuberosity to medial epicondyl of femur.
  Sessions: Total 8 sessions will be given 2 sessions per week for 4 weeks.
  Other Names: Group A
  Arms: Dry Needling
Other: Soft Tissue Mobilization — Baseline Treatment: Hot pack will be applied for 15 minutes on Hamstrings and lower back and transcutaneous electrical nerve stimulation (TENS) at lower back for warm up and pain relief to both groups. Then spinal mobilization (Poster lateral glide) of grade 1 and 2 (3 sets of 6 repetitions) i.e. within the spine resistance.
  Soft Tissue Mobilization will be given to Group B along with Baseline treatment.
  Subject will be in prone lying position with knee bent at 30 to 60 degrees. Soft tissue mobilization will be applied on hamstring muscle through Graston technique. Massage cream will be applied on hamstring muscle and Graston Instrument will be rubbed from gluteal line to politeal fossa 30 times for 60 seconds.
  Sessions: Total 8 sessions will be given 2 sessions per week for 4 weeks.
  Other Names: Group B
  Arms: Soft Tissue Mobilization

SUMMARY:
The hamstring tightness is considered as the inability to achieve knee extension greater than 160 degrees while hip is flexed at 90 degrees. When low back pain (LBP) persists for 12 weeks or longer, it is termed as chronic low back pain. The objective of study is to see the effect of dry needling versus soft tissue mobilization on hamstring muscle on pain, range of motion and functionality in patients with chronic low back pain.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted at Hameed Latif Medical Centre through non probability convenient sampling technique on 30 subjects which will be divided into two groups' 15 subjects in group A and 15 subjects in group B through computer generated software for Randomization. Both groups will be conventional therapy and spinal mobilization (posterior anterior glide) of grade 1 and 2 (3 sets of 6 repetitions) as baseline treatment. Group A was will be dry needling and Group B will be Soft Tissue Mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Reduction in active knee extension test >25
* Current back pain between 4 to 6 on Numeric Pain Rating scale
* Low back pain for at least 12weeks0r 6 months

Exclusion Criteria:

* Subjects using anticoagulants and having vascular diseases
* Subjects with needle phobia and allergic to metals
* Subjects with cognitive impairment
* History of fracture in lumbar region
* History of systemic diseases e.g. cancer or systemic joint pathologies
* History of congestive heart failure in past 24 months
* Subjects have used medications like narcotics or Muscle relaxants 30 days before enrolment into study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  Numeric Pain Rating Scale (NPRS) was used to measure low back pain. NPRS consists of 11 points, which range from 0= no pain, 1-4= mild pain, 4-7= moderate pain 7-10= severe pain . Researchers states that NPRS shows High test to re test reliability (ICC 0.96) in elderly populations with musculoskeletal disorders without having cognitive dysfunction.
Oswestry Disability index (Urdu) | 4 weeks
  The Oswestry Disability index (ODI) consists of 10 patient- completed questions in which the response options are presented as 6-point Likert scales. Scores range from 0% (no disability) to 100% (most severe disability).
Inclinometer | 4 weeks
  It was used to measure range of motion of low back. An instrument for measuring angles is an inclinometer. A sensor is housed in the housing of an inclinometer. The sensor measures the housing's tilt and is sensitive to gravity. After that, the angle is shown on a dial or digital display.
Active Knee Extension Test | 4 Week
  The most effective way to exclude the hamstring muscle's extensibility range, with the hip fixed at a 90-degree angle and precise instrument placement, is to perform the active knee extension test. This technique provides accurate measures of hamstring length and extensibility when used in a supine 90/90 position. Both a normal goniometer and an electrogoniometer were used to measure the amount of extension. Whether hamstring tightness contributes to mechanical low back pain can be inferred from this result.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Hameed Latif Medical Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No